CLINICAL TRIAL: NCT06754228
Title: Acute Immune Modulation by Probiotic Strain Bacillus Coagulans JBI-YZ6.3 (BC4U)
Brief Title: Acute Immune Modulation by Probiotic Strain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Collaborators: Jeneil Biotech Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 187-008
Record Dates: First submitted 2024-11-12; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Immune Surveillance

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, escalating dose, cross-over study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group A (Experimental): Crossover study: Participants will be consuming placebo on the first clinic visit, a low dose of the probiotic on the second clinic visit, a medium dose of the probiotic on the third clinic visit, and a high dose of the probiotic on the fourth clinic visit. Each clinic visit is separated by at least 1 week wash-out period.
  Interventions: Dietary Supplement: Probiotic Agent

INTERVENTIONS:
Dietary Supplement: Probiotic Agent — Bacillus coagulans JBI-YZ6.3 (BC4U)
Dietary Supplement: Probiotic Agent — An escalating dose cross-over design: Participants are fed 0 mg, 100 mg, 200 mg, and 400 mg on different clinic visits.

SUMMARY:
Clinical proof-of-concept study, comparing the acute immune impacts of 3 doses of a probiotic strain to a placebo. This study involves twenty-four participants, composed of healthy adults, who will be taking a placebo and 3 different doses of the probiotic at different times. Testing for immune status and cytokine levels will be conducted to determine the acute impact of the probiotic on immune function when compared to a placebo.

DETAILED DESCRIPTION:
Clinical proof-of-concept study comparing the acute immune effects of 3 doses of a probiotic compared to a placebo. The probiotic strain is characterized as Bacillus coagulans JBI-YZ6.3 (BC4U).

24 subjects will participate in a placebo-controlled, escalating dose, cross-over study design, wherein they will be taking placebo, dose 1, dose 2, and dose 3, each separated by a 1-week washout period.

Blood samples are taken 1 hour after participants arrive; the dose is then administered. Samples are taken 1 hour, 2 hours, and 3 hours following administration.

A series of immune panels will be used to determine the acute impacts on immune surveillance, immune cell activation status, immune cell priming, and cytokine profiles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-75 years (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with study procedures, including:

  * Maintaining a consistent diet and lifestyle routine throughout the study,
  * Consistent habit of bland breakfasts on days of clinic visits,
  * Abstaining from exercising and nutritional supplements on the morning of a study visit,
  * Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
  * Abstaining from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/ life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Pregnant, nursing, or trying to become pregnant;
* Known food allergies related to ingredients in active test product or placebo.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Immune communication | 3 hours
  Changes in serum cytokine levels

SECONDARY OUTCOMES:
Immune surveillance and alertness | 3 hours
  Changes in immune cell trafficking and status of immune cell alertness, ie. the changes in immune cell populations and activation status following consumption:
  Numbers of CD3- CD56+ NK cells in blood Numbers of CD3+ CD56+ NKT cells in blood Numbers of CD3+ CD56- T cells in blood Numbers of cells positive for CD25 Numbers of cells positive for CD69

OTHER OUTCOMES:
Immune responsiveness | 3 hours
  Ex vivo immune challenges, documenting the capabilities of anti-bacterial and anti-viral immune responses:
  Cytokine levels in 24-hour culture supernatants of ex vivo immune cell cultures in unchallenged cultures Cytokine levels in 24-hour culture supernatants of ex vivo immune cell cultures in lipopolysaccharide-inflamed cultures Cytokine levels in 24-hour culture supernatants of ex vivo immune cell cultures in Poly I:C challenged cultures

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No